CLINICAL TRIAL: NCT00714064
Title: PneuMum: A Randomised Controlled Trial of Pneumococcal Polysaccharide Vaccination for Aboriginal and Torres Strait Islander Mothers to Protect Their Babies From Ear Disease
Brief Title: PneuMum: Pneumococcal Vaccination of Australian Indigenous Mothers
Acronym: PneuMum
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Ross Andrews, Professor, Menzies School of Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHMRC 490320; NHMRC 350499
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Middle Ear Effusion; Tympanic Membrane Perforation; Acute Otitis Media; Pneumococcal Infections
MeSH Terms: conditions — Otitis Media with Effusion; Tympanic Membrane Perforation; Otitis Media; Pneumococcal Infections | interventions — Pentetic Acid; Pneumococcal Vaccines; Boostrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 23vPPV in Pregnancy (Active Comparator)
  Interventions: Biological: 23vPPV, dTpa (Pneumovax, Boostrix)
- 23vPPV at Birth (Active Comparator)
  Interventions: Biological: 23vPPV, dTpa (Pneumovax, Boostrix)
- Control (Other): Control
  Interventions: Biological: 23vPPV, dTpa (Pneumovax, Boostrix)

INTERVENTIONS:
Biological: 23vPPV, dTpa (Pneumovax, Boostrix) — Group A will receive 23vPPV during 3rd trimester and dTpa at delivery
  Other Names: Pneumovax, Boostrix
  Arms: 23vPPV in Pregnancy
Biological: 23vPPV, dTpa (Pneumovax, Boostrix) — Group B will receive 23vPPV at delivery and dTpa 7 months following delivery
  Other Names: Pneumovax, Boostrix
  Arms: 23vPPV at Birth
Biological: 23vPPV, dTpa (Pneumovax, Boostrix) — Group C will receive dTpa at delivery and 23vPPV 7 months following delivery
  Other Names: Pneumovax, Boostrix
  Arms: Control

SUMMARY:
PneuMum is a randomised controlled trial that aims to find out if pneumococcal vaccination for Australian Indigenous mothers, in the last few months of pregnancy or at delivery, can prevent ear disease in infants. Mothers will receive the 23 valent pneumococcal polysaccharide vaccine (23vPPV) either: a) during the third trimester of pregnancy; b) soon after child birth; or c) seven months after child birth (control group). The adult diphtheria, tetanus and acellular pertussis vaccine (dTpa) will be used as the control vaccine for the birth dose.

The study aims to recruit 210 Indigenous women aged 17-39 years who have an uncomplicated pregnancy. Following recruitment, subjects will be randomly assigned to one of the three groups.

Each mother and infant will be followed from pregnancy until the baby is seven months of age. All routinely recommended vaccinations on the standard vaccination schedule will continue to be offered by the subject's vaccine provider in accordance with current clinical practice.

The primary outcome will be prevalence of middle ear disease at seven months of age, defined as middle ear effusion or tympanic membrane perforation or acute otitis media. Pneumatic otoscopy, video-otoscopy and tympanometry will be used in the ear examinations. The primary analyses will be a direct comparison of the proportion of infants in the control group who have nasopharyngeal carriage of one or more vaccine type pneumococci at seven months of age compared to infants in each of the other two groups. A similar comparison of the proportion with middle ear disease will be undertaken between the control group and the respective intervention group.

DETAILED DESCRIPTION:
PneuMum is a randomised controlled trial that aims to find out if pneumococcal vaccination for Australian Indigenous mothers, in the last few months of pregnancy or at delivery, can prevent ear disease in infants. Two vaccines will be used in this trial:

* The 23 valent pneumococcal polysaccharide vaccine (23vPPV), is currently recommended for all Indigenous people in the Northern Territory from 15 years of age but uptake among women of child-bearing age has been low.
* Adult diphtheria, tetanus and acellular pertussis vaccine (dTPa) will be used as the control vaccine. This vaccine is recommended for all new parents who have not previously been immunised but is not currently funded so would normally need to be purchased on prescription through a pharmacist.

Rationale

Indigenous children experience the highest rates of acute and chronic ear infections in the world, resulting in permanent ear damage, hearing loss and educational disadvantage. These infections are mainly bacterial. Streptococcus pneumoniae (pneumococcus) is the predominant pathogen. Pneumococcal colonisation and infection begins within days of birth, months before any potential immunological protection from infant pneumococcal conjugate vaccine may be expected. New strategies are needed to eliminate, or at least delay, this early-onset pneumococcal colonisation.

Maternal vaccination with the 23 valent pneumococcal polysaccharide vaccine (23vPPV) during pregnancy or at delivery is one strategy that may protect newborn infants through mechanisms such as transplacental antibody transfer, increased secretory antibody in breast milk, and/or by reducing nasopharyngeal carriage (and transmission to the infant) of maternal pneumococci. Previous small studies using this strategy have been encouraging, but there have been no studies properly evaluating nasopharyngeal carriage or disease endpoints in infants.

Methods

We aim to recruit 210 Indigenous women aged 17-39 years who have an uncomplicated pregnancy. Following recruitment, subjects will be randomly assigned to one of three groups:

* Group A will receive 23vPPV in the last few months of pregnancy
* Group B will receive 23vPPV soon after childbirth
* Group C will receive 23vPPV seven months after childbirth (the control group).

Women in Groups A and C will receive dTpa soon after childbirth (to conceal the intervention groups), whereas women in Group C will be offered dTpa seven months after childbirth (end of the observation period).

Study participants will be visited at least five times:

1. During the last few months of pregnancy (30-36 weeks gestation)

   - The group of mothers receiving 23vPPV at this visit will also have a pre-vaccination blood sample collected
2. At Royal Darwin Hospital when the baby is born

   * Each mother will receive either 23vPPV or dTpa depending on their allocation
   * Each mother will have a pre-vaccination blood sample, cord blood sample, a nasopharyngeal swab and a sample of expressed breast milk taken
3. When the baby is one month old

   - Each baby will have their ears checked utilising pneumatic otoscopy, video-otoscopy and tympanometry. A nasopharyngeal swab will be taken. A swab will also be taken of any discharge from the baby's ear/s. Mothers will be asked for sample of expressed breast milk and a post vaccine maternal blood sample will be collected.
4. When the baby is two months old

   - The same checks and samples as the previous month with the exception of maternal blood sample unless this has not previously been collected.
5. When the baby is seven months old - Each mother and baby will have the same checks and samples as per the two month visit. Babies will also have a sample taken of their blood. Mothers who have not yet had 23vPPV will be offered that vaccine as will those who have not yet had dTpa.

Primary Outcome

The primary outcomes will be:1)prevalence of middle ear disease at seven months of age; and 2)prevalence of nasopharyngeal carriage of vaccine type (23vPPV) pneumococci. The primary analyses will be a direct comparison of the proportion of infants in the control group (Group C) who have nasopharyngeal carriage of vaccine type pneumococci at seven months of age compared to infants in each of the other two groups and a similar comparison of the proportion with middle ear disease.

ELIGIBILITY:
Inclusion Criteria:

* Singleton uncomplicated pregnancy
* Reside in Darwin, the Tiwi Islands, or other remote community where consent has been obtained
* Intends to deliver child at the Royal Darwin Hospital or other designated hospital where consent has been obtained
* Has given informed consent to participate

Exclusion Criteria:

* Had 23vPPV within the previous three years
* Had a previous dose of dTpa
* Intends to leave the study area during the follow-up period
* HIV positive
* History of severe allergy, uncontrolled asthma or splenectomy

Ages: 17 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 227 (Actual)
Dates: Start 2006-06; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of middle ear disease, defined as middle ear effusion or tympanic membrane perforation or acute otitis media | at seven months of age
Nasopharyngeal carriage of vaccine type pneumococci | at seven months of age

SECONDARY OUTCOMES:
Prevalence of middle ear disease | at one month of age
Nasopharyngeal carriage of vaccine type pneumococci | at one month of age
Prevalence of middle ear disease | at two months of age
Nasopharyngeal carriage of vaccine type pneumococci | at two months of age
Relationship of maternal pneumococcal carriage, maternal anti-pneumococcal antibody levels, cord blood antibody levels and breast milk antibody levels to infant carriage and middle ear disease | at one, two and seven months of age
Impact of each maternal vaccination strategy on breast milk antibody levels to serotypes contained in the vaccine | at seven months
Impact of each maternal vaccination strategy on breast milk antibody avidity (to four selected serotypes) | at seven months
Impact of each maternal vaccination strategy on maternal antibody response to antepartum or postpartum 23vPPV | at seven months
Impact of each maternal vaccination strategy on infant anti-pneumococcal antibody levels (following the 3rd recommended dose of 7vPCV) | at seven months of age

CONTACTS AND LOCATIONS:
Overall Officials: Ross M Andrews, PhD, Principal Investigator — Menzies School of Health Research; Jonathan R Carapetis, PhD, Principal Investigator — Menzies School of Health Research; Amanda J Leach, PhD, Principal Investigator — Menzies School of Health Research; Peter S Morris, PhD, Principal Investigator — Menzies School of Health Research; Edward K Mulholland, DM, Principal Investigator — The Univeristy of Melbourne and Murdoch Childrens Research Institute; Paul J Torzillo, MBBS, Principal Investigator — Royal Prince Alfred Hospital, Sydney; Mimi LK Tang, PhD, Principal Investigator — Royal Children's Hospital
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- [Derived] Martinovich KM, Seppanen EJ, Bleakley AS, Clark SL, Andrews RM, Richmond PC, Binks MJ, Thornton RB, Kirkham LS. Evidence of maternal transfer of antigen-specific antibodies in serum and breast milk to infants at high-risk of S. pneumoniae and H. influenzae disease. Front Immunol. 2022 Sep 21;13:1005344. doi: 10.3389/fimmu.2022.1005344. eCollection 2022. PMID 36211411
- [Derived] Binks MJ, Moberley SA, Balloch A, Leach AJ, Nelson S, Hare KM, Wilson C, Nelson J, Morris PS, Ware RS, Tang MLK, Torzillo PJ, Carapetis JR, Mulholland K, Andrews RM. Impact of the 23-valent pneumococcal polysaccharide vaccination in pregnancy against infant acute lower respiratory infections in the Northern Territory of Australia. Pneumonia (Nathan). 2018 Dec 25;10:13. doi: 10.1186/s41479-018-0057-2. eCollection 2018. PMID 30603376
- [Derived] Binks MJ, Moberley SA, Balloch A, Leach AJ, Nelson S, Hare KM, Wilson C, Morris PS, Nelson J, Chatfield MD, Tang ML, Torzillo P, Carapetis JR, Mulholland EK, Andrews RM. PneuMum: Impact from a randomised controlled trial of maternal 23-valent pneumococcal polysaccharide vaccination on middle ear disease amongst Indigenous infants, Northern Territory, Australia. Vaccine. 2015 Nov 27;33(48):6579-87. doi: 10.1016/j.vaccine.2015.10.101. Epub 2015 Oct 31. PMID 26529076
- See also: Previous Registration History - through University of Melbourne — http://www.clinicaltrials.gov/ct2/show/NCT00310349?term=Pneumum+AND+Australia&rank=1